CLINICAL TRIAL: NCT00453245
Title: Study of the Molecular Basis of the Growth Axis Among Short Stature Children
Brief Title: Molecular Basis of the Growth Axis in Short Stature
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Other Study IDs: 920040018
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2007-03-28 (Estimated); Status verified 2004-01

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To examine the clinical genetic and biochemical characteristics of children with growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patient with growth hormone deficiency

Ages: 1 Year to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-01; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yardena T Rakover, MD, Principal Investigator — haemek medical center
Locations (1):
- Haemek Medical Center, Afula, Israel